CLINICAL TRIAL: NCT05904626
Title: A Multi-center, Double-Blind, Randomized, Two-Arm, Parallel-Group, Placebo Controlled Basket Study to Assess the Safety of ELGN-2112 in Preterm Infants Born Under 26 Weeks GA and IUGR Infants Born 26-32 Weeks GA
Brief Title: Assess the Safety of ELGN-2112 in Preterm Infants Born Under 26 Weeks GA and IUGR Infants Born 26-32 Weeks GA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Elgan Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FIT-05
Record Dates: First submitted 2023-03-30; First posted 2023-06-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Intestinal Malabsorption
MeSH Terms: conditions — Malabsorption Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ELGN-2112 Human insulin [rDNA] (Active Comparator)
  Interventions: Drug: ELGN-2112
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ELGN-2112 — To compare the safety of treatment with ELGN-2112 to placebo in preterm infants born less than 26 weeks GA and IUGR infants<3rd percentile* born at 26-32 weeks GA.
  Arms: ELGN-2112 Human insulin [rDNA]
Drug: Placebo — A placebo formulation consisting of the same inactive ingredients as ELGN-2112.
  Arms: Placebo

SUMMARY:
To compare the safety of treatment with ELGN-2112 to placebo in preterm infants born less than 26 weeks GA and IUGR infants<3rd percentile* born at 26-32 weeks GA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female preterm infant born less than 26 weeks GA or Intra-Uterine Growth Restricted infants born between 26+0 to 31+6 GA.
* Birth weight ≥ 450g
* Singleton or twin birth

Exclusion Criteria:

N/A

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Compare the safety of treatment with ELGN-2112 to placebo in preterm infants born less than 26 weeks GA | Five days from birth until 42 days
  Safety will be assessed by capturing of adverse events (AEs) during the treatment period.
Compare the safety of treatment with ELGN-2112 to placebo in preterm infants born IUGR infants<3rd percentile* born at 26-32 weeks GA. | Five days from birth until 42 days
  Safety will be assessed by capturing of adverse events (AEs) during the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Miki Olshansky, Study Director — Elgan Pharma Ltd.